CLINICAL TRIAL: NCT03177876
Title: Schneiderian Membrane Elevation and Augmentation With Hydroxyapatite Nano Particles [ Nano Streams ] Versus Graft Less Tenting Technique With Simultaneous Implant Placement: Randomized Clinical Trial
Brief Title: Sinus Lift With Hydroxyapatite Nano Particles Versus Tenting Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hossam Khaled Shehata Faraag, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebc.cairo university
Record Dates: First submitted 2017-05-19; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Maxillary Sinus Lift
Keywords: tenting Hydroxyapetite nano particles implant immediate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sinus lift implant placement Hydroxyapatite Nano particles (Experimental): shneiderian membrane elevation and augmentation with Hydroxyapatite Nano particles [Nanostreams] with simultaneous implant placement
  Interventions: Procedure: sinus lift implant placement Hydroxyapatite Nano particles
- sinus lift implant placement tenting (Active Comparator): shneiderian membrane elevation and augmentation with graft less tenting technique with simultaneous implant placement
  Interventions: Procedure: sinus lift implant placement tenting

INTERVENTIONS:
Procedure: sinus lift implant placement Hydroxyapatite Nano particles — shneiderian membrane elevation and augmentation with Hydroxyapatite Nano particles with simultaneous implant placement
  Arms: sinus lift implant placement Hydroxyapatite Nano particles
Procedure: sinus lift implant placement tenting — shneiderian membrane elevation and augmentation with graft less tenting technique with simultaneous implant placement
  Arms: sinus lift implant placement tenting

SUMMARY:
twenty recruited patients indicated for sinus augmentation and immediate implant placement will be divided into two groups (10 in each of the two groups), to compare bone formation and implant stability after shneiderian membrane elevation and augmentation with Hydroxyapatite Nano particles [Nanostreams] or augmentation with graft less tenting technique with simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic maxilla and pneumatization of the maxillary sinus with residual bone height at least 5mm of residual ridge as per MISCH criteria
* Both sexes

Exclusion Criteria:

* Sinus pathology
* Heavy smokers more than 20 cigarettes per day
* Patients with systemic disease that may affect normal healing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 7 days post operative
  evaluation of post operative complications in terms of pain and edema using patient pain chart

SECONDARY OUTCOMES:
implant stability | will be measured intra-operative after implant insertion and will be measured one more time 6 months after the first operation at the time of implant exposure
  measurement of the implant stability using osstell device
height of bone gain or loss around the implant | 6 months post operative
  two cone beam CT will be taken for the patients, one immediate post operative and the other 6 months post-operative then the amount of bone gained or loss will be assessed by superimposing the same section in the two cone beam CT

IPD SHARING:
Plan to Share IPD: Yes